CLINICAL TRIAL: NCT00484653
Title: Identification and Impact of Vaginal Flora Anomalies Among Pregnant Woman
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2007/07
Record Dates: First submitted 2007-06-08; First posted 2007-06-11 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Vaginosis, Bacterial
Keywords: To achieve a quality and quantitative molecular biology assay for vaginal flora abnormalities
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — Vaginal Smears

INTERVENTIONS:
Procedure: cervical smear — biological analysis

SUMMARY:
This is a prospective multicentric study including six clinical units of Gynecology and Obstetrics (5 public health hospital and one private team), one research team in clinical microbiology and one Center of Clinical investigation (CIC).

There is a correlation between premature delivery and bacterial vaginosis. So, the anomalies of vaginal flora are a potential target for the campaign against prematurity.

The main objective of this study is to achieve an objective and reproducible technique of identification and quantification by molecular biology of lactobacilla and all the other micro-organisms involved in vaginal flora anomalies.

The secondary objectives are the exhaustive culture of bacteria, the characterisation of intermediate vaginal flora and bacterial vaginosis among pregnant woman by PCR targeting the ribosomic ADN 16S coupled with clonage techniques.

The number of patient to include is 1000 (time of inclusions: 24 months). The vaginal smears will be realized until 32 weeks of gestation (Max: 3 taking of vaginal smears by patient).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients aged more than 18 years and more than 14 weeks of gestation but less than 28 weeks.
* Multiple pregnancy won't be included.
* Patient with a risk of premature delivery with a short cervix or a cervix measured at less than 25 mm (measure done by vaginal ultrasound of the cervix).
* Or patient with a past of premature delivery and/or of late abortion.
* Symptomatic or asymptomatic patient.
* Patients consulting for pregnancy follow up or hospitalized in a unit of Gynecology and Obstetrics involved in the study.
* social security cover
* written informed consent

Exclusion Criteria:

* antecedents : treated hypertension, Foetal malformation, APLS known, diabetes, renal disease, SLE
* treated with antibiotics the inclusion's day
* dropping consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Actual)
Dates: Start 2007-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
identification and quantification by molecular biology of lactobacilla and all the other micro-organisms involved in vaginal flora anomalies | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Florence BRETELLE, PU-PH, Principal Investigator — Assistance Publique Hôpitaux de Marseille
Locations (6):
- France (6):
  - CHU Antoine BECLERE, Clamart
  - Hôpital Saint Joseph, Marseille
  - Hôpital Nord-OB/GYN Department, Marseille
  - Hôpital de la Conception, Marseille
  - Centre Hospitalier Poissy-Saint-Germain, Poissy
  - Centre médicochirurgical et obstétrical, Schiltigheim

REFERENCES:
- [Derived] Bretelle F, Rozenberg P, Pascal A, Favre R, Bohec C, Loundou A, Senat MV, Aissi G, Lesavre N, Brunet J, Heckenroth H, Luton D, Raoult D, Fenollar F; Groupe de Recherche en Obstetrique Gynecologie. High Atopobium vaginae and Gardnerella vaginalis vaginal loads are associated with preterm birth. Clin Infect Dis. 2015 Mar 15;60(6):860-7. doi: 10.1093/cid/ciu966. Epub 2014 Dec 1. PMID 25452591
- [Derived] Menard JP, Fenollar F, Raoult D, Boubli L, Bretelle F. Self-collected vaginal swabs for the quantitative real-time polymerase chain reaction assay of Atopobium vaginae and Gardnerella vaginalis and the diagnosis of bacterial vaginosis. Eur J Clin Microbiol Infect Dis. 2012 Apr;31(4):513-8. doi: 10.1007/s10096-011-1341-8. Epub 2011 Jul 26. PMID 21789604
- [Derived] Menard JP, Mazouni C, Salem-Cherif I, Fenollar F, Raoult D, Boubli L, Gamerre M, Bretelle F. High vaginal concentrations of Atopobium vaginae and Gardnerella vaginalis in women undergoing preterm labor. Obstet Gynecol. 2010 Jan;115(1):134-140. doi: 10.1097/AOG.0b013e3181c391d7. PMID 20027045